CLINICAL TRIAL: NCT06858787
Title: The Validity of a Continuous Glucose Monitor in Diagnosing Gestational Diabetes: A Pilot Study
Brief Title: Validating CGM for GDM
Acronym: VALID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Angela Bianco, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-25-00172
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Individuals receiving prenatal care at Mount Sinai Hospital (Experimental): Women receiving prenatal care at Mount Sinai Hospital to have 10-day application of continuous glucose monitor
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — Device is a remote sensor applied to the upper extremity that continuously samples glucose of interstitial fluid and uploading results to a mobile application.

SUMMARY:
This is a prospective pilot study to assess the validity of using a continuous glucose monitor (CGM) in diagnosing gestational diabetes mellitus (GDM). Pregnant individuals between the ages of 18-50 years old receiving prenatal care at Mount Sinai Hospital (e..g, E-Level clinic and Faculty Practice Associates) will be enrolled. Potential participants will be approached during their prenatal care appointments. Participants will complete an informed consent form for the study during their standard-of-care prenatal appointments at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Singleton pregnancy between 24-32 weeks gestational age
* Prenatal care and delivery at Mount Sinai Hospital

Exclusion Criteria:

* Multiple fetal gestation
* Preexisting diabetes
* Concurrent use of steroids
* Anomalous fetus
* Insufficient prenatal care (identified as missing half the recommended visits or establishing care after 20 weeks gestation)
* Unable to tolerate oral glucose test

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Blood glucose from CGM | 10 days from sensor application to completion of testing
  Blood glucose aggregate values from Dexcom G7 continuous glucose monitor (CGM)
Glucose Tolerance Test (GTT) values | 1 hour and 3 hours
  1-hour GTT values and 3-hour GTT values
  The glucose tolerance test is a lab test to check how the body moves sugar from the blood into tissues like muscle and fat. The test is used as standard of care to diagnose gestational diabetes.
Postpartum blood glucose | 4 hours after childbirth
  A blood sugar test measures the amount of a sugar called glucose in a sample of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bianco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai South Nassau, Oceanside, New York

IPD SHARING:
Plan to Share IPD: No